CLINICAL TRIAL: NCT03997214
Title: The Impact of Inspiratory Muscle Strength Training on Weaning Parameters Among Ventilator-dependent Patients
Brief Title: The Impact of Inspiratory Muscle Strength Training
Acronym: IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fooyin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 108001
Record Dates: First submitted 2019-06-04; First posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-05

CONDITIONS: Ventilator Dependency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): as usual care
- experimental group (Experimental): The intervention of inspiratory muscle strength training
  Interventions: Device: inspiratory muscle strength training

INTERVENTIONS:
Device: inspiratory muscle strength training — The experimental group received the intervention of inspiratory muscles training 5times/week for 6 weeks, 5days/ per cycle; the patients stayed in the semi-recumbent position, recorded the initial/first measurement of MIP. The trigger sensitivity was adjusted to 10% of the first recorded MIP at the start of training, then reducing the ventilator trigger sensitivity and training duration weekly.
  Arms: experimental group

SUMMARY:
The study is a pre-post test with quasi experimental design. Forty-two intubated-adults who had been mechanically ventilated for more than 21 days were selected on the basis of inclusion criteria in respiratory care ward. These patients were classified equally into study group and control group. The experimental group received the intervention of respiratory muscles training 5 times/ a week for 6 weeks. The control group received normal care. The intervention was adjusted trigger sensitivity to 10% of the first recorded Maximal Inspiratory Pressure at the start of training, then increased the ventilator trigger sensitivity and training duration weekly. The largest of ventilator trigger sensitivity is not over 40% of the initial Maximal Inspiratory Pressure and the timing of training duration is no longer than 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age >20y/o
* Vital signs stable
* MIP <20cmH2O
* Ventilator FiO2<40%, PEEP <8
* Ventilator mode:PSV or SIMV

Exclusion Criteria:

* Patient or family refuse

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure | 7 weeks
  a measure of the strength of inspiratory muscles, measurement by cmH2O.
Tidal volume | 7 weeks
  the volume of air that is transported into and out of the lungs with each respiratory cycle, measurement by mL per inspiration
Minute ventilation volume | 7 weeks
  the quantity of air moved into and out of the lungs in a minute, measurement by l.min
Rapid shallow breathing index | 7 weeks
  the ratio of respiratory frequency to tidal volume (f/VT)
Oxygenation index. | 7 weeks
  Oxygenation index OI = FiO2 x 100 x M AP/PaO2, where FiO2 is the fraction of inspired oxygen, MAP is the mean airway pressure, and PaO2 is the partial pressure of oxygen in arterial blood, calculated at the end of the first day of standardized preoperative stabilization

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Yun Chang, Ph.D, Principal Investigator — Fooyin
Locations (1):
- Shinghou Hospital, Kaohsiung City, Fengshan, Taiwan

IPD SHARING:
Plan to Share IPD: No